CLINICAL TRIAL: NCT00778687
Title: Effects of Liver Transplantation on the Heart Rate Variability in Patients With End-Stage Liver Disease
Brief Title: Heart Rate Variability Change After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200809046R
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cirrhotic cardiomyopathy describes a hyperdynamic state with the presentation of high cardiac output and low systemic vascular resistance. And the latent heart failure becomes obvious under physiologic and pharmacologic stress. The goal of our study is to assess the effects of liver transplantation on the heart rate variability in patients with end stage liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-70y/o receiving liver transplantation

Exclusion Criteria:

* History of cardiovascular disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end stage liver disease undergoing liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Multiscale entropy | 6 months
  Multiscale entropy was measured at nine time points: 1. preoperative, 2. postoperative day 1, 3. postoperative day 2, 4. postoperative day 3, 5. postoperative day 4, 6. postoperative day 7, 7. postoperative day 14, 8. postoperative 3 months, 9. postoperative 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Genovesi S, Prata Pizzala DM, Pozzi M, Ratti L, Milanese M, Pieruzzi F, Vincenti A, Stella A, Mancia G, Stramba-Badiale M. QT interval prolongation and decreased heart rate variability in cirrhotic patients: relevance of hepatic venous pressure gradient and serum calcium. Clin Sci (Lond). 2009 May 14;116(12):851-9. doi: 10.1042/CS20080325. PMID 19076059